CLINICAL TRIAL: NCT03453957
Title: Therapeutic Alliance Tensions and Repair in Psychotherapy Practices: A Psychotherapy Practice Research Network (PPRNet) Study
Brief Title: Therapeutic Alliance Tensions and Repair in Psychotherapy Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Giorgio A. Tasca, Associate Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 363733
Record Dates: First submitted 2018-02-16; First posted 2018-03-05 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Psychotherapy; Therapeutic Alliance
Keywords: Practice based research

STUDY DESIGN:
Intervention Model Description: This will be a 2-arm, parallel, prospective, single-blind cluster RCT with 1-1 allocation comparing: (a) therapists who receive the professional development intervention to identify and repair alliance tensions at the study outset versus (b) therapists who receive the intervention after participation is complete (no training control). Therapists will be randomized to study condition and patients will be clustered within therapists. Randomization will control for: (a) the effect of therapist variables (age, gender, theoretical orientation, experience, differing initial skill level) on competence, therapeutic alliance, or patient outcomes; (b) potential biases caused by pre-treatment patient variables (symptom severity, co-morbidity, chronicity, psychoactive medications); and (c) treatment or study factors (e.g. frequency of sessions, time to complete the study sessions, treatment received after the study sessions). Patients will be blind to therapist study arm allocation.
Who Masked: Participant
Masking Description: Participating therapists will be aware of their group (Professional development training vs no training control); however, their participating patient/clients will not know which experimental group their therapists belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Professional Development Program (Experimental): Therapists who participate in workshops and consultation sessions with study trainers during study-related therapy sessions and their participating patients/clients.
  Interventions: Other: Professional development program
- Control (No Intervention): Therapists who did not participate in workshops and consultations sessions while engaging in study-related therapy sessions and their participating patients/clients.

INTERVENTIONS:
Other: Professional development program — Professional development program consists of training including workshops and consultation sessions to enhance therapists ability to detect and repair alliance ruptures in active community based psychotherapy.
  Arms: Professional Development Program

SUMMARY:
This study evaluates a professional development program intended to improve the relationship or alliance between therapists and patients/clients who are receiving psychotherapy in the community. Half of the participating therapists will receive training to detect and improve alliance with new patients while half will not. The professional development training is expected to improve therapists effectiveness in identifying and correcting alliance tensions which will, in turn, improve therapeutic outcomes for patients/clients.

DETAILED DESCRIPTION:
Psychotherapy is the treatment of choice for many mental disorders, yet there is a gap between research and practice. Research indicates that: the therapist-patient alliance is important to reduce patient symptoms, alliance tensions are detrimental to patients, and those therapists who identify and repair alliance tensions can improve patient outcomes. In this study we will use state of the art research to train community-based therapists in evidence-based interventions to identify and repair alliance tensions. Trained therapists and their patients will be compared to therapists who provide usual care to their patients. Improvement in therapists' skills in identifying and repairing alliance tensions and how this is associated with better patient mental health outcomes will be measured. Trained therapists will be interviewed to identify the best ways of improving the training and disseminating the findings to psychotherapists across Canada. Research to improve practicing therapists' ability to identify and repair therapeutic alliance tensions will result in better mental health outcomes for patients.

ELIGIBILITY:
Therapist

Inclusion Criteria:

* regulated health professional
* in good standing with a Canadian provincial regulatory college
* scope of practice includes psychotherapy
* ability to add 3 or more new, English speaking clients to caseload over 6 to 9 months
* ability to obtain timely permission to conduct research from therapist's employing institution or health group when applicable

Exclusion Criteria:

* none

Patient/Client

Inclusion Criteria:

* 18 years of age or older
* will participate in psychotherapy sessions in English
* will see the study-affiliated therapist for a minimum of 6 sessions in the next 6 months

Exclusion Criteria:

* already seeing another therapist
* diagnosed with a neurocognitive disorder
* diagnosed with a psychotic disorder
* expressed suicidal behaviour in the past six months as assessed by their participating therapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
Mean tension resolution rating scale | 6 therapy sessions over 6 weeks up to 6 months depending on the frequency of therapy
  The Rupture Resolution Rating System (3RS) is an observer-based measure to identify alliance tensions and resolution processes. Independent blind reliable trained judges will rate video recordings of 6 psychotherapy session recorded with participating clients. A mean tension score will be assigned per client which will be the average of the 6 session scores.
  score ranges from 1 (withdrawal/confrontation rupture(s) did not occur; not significant for the alliance) to 5 (withdrawal/confrontation rupture(s) occurred; significant for the alliance).

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 7-item scale (GAD-7) change from baseline | baseline and end of 6 therapy sessions, 6 weeks to 6 months depending on the frequency of therapy
  Self-report measurement of severity of anxiety using the GAD-7 scale. A change in anxiety scores will be assess following 6 therapy session with data collected before therapy(baseline) and again after all 6 sessions of therapy have been completed. Scores range from 0 (low anxiety) to 27 (high anxiety) with scores over 10 being of clinical significance.
Patient Health Questionnaire 9-item scale (PHQ-9) change from baseline | baseline and end of 6 therapy sessions, 6 weeks to 6 months depending on the frequency of therapy
  Self-report measurement of depression symptoms using the PHQ-9 scale. A change in depression symptom scores will be assess following 6 therapy session with data collected before therapy and again after all 6 sessions of therapy have been completed. Scores range from 0 (low) to 27 (high) with scores over 10 being of clinical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Tasca, Ph.D., Principal Investigator — University of Ottawa
Locations (2):
- Canada (2):
  - University of Ottawa, Ottawa, Ontario
  - Mt. Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PPRNet website including study-related information and publications — http://www.pprnet.ca